CLINICAL TRIAL: NCT01373541
Title: Effect of InFat™ Product on Stool Biochemistry and Stool Characteristics in Formula-fed Term Infants in China: a Double Blind, Multi-center, Randomized, Controlled Trial
Brief Title: Effect of InFat™ Product on Stool Biochemistry and Stool Characteristics in Formula-fed Term Infants in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enzymotec (Industry)
Collaborators: Biostime, Inc. (Guangzhou) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: InFat_003
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2012-01

CONDITIONS: Health Behavior; Personal Satisfaction
MeSH Terms: conditions — Health Behavior; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- InFat group (Active Comparator): Infant formula with structured triglycerides (high palmitic acid content at the sn-2 position)
  Interventions: Other: InFat™ based infant formula
- Control group (Active Comparator): Infant formula with standard vegetable blend (low palmitic acid content at the sn-2 position)
  Interventions: Other: Standard vegetable oil based infant formula
- Referance group (No Intervention): Human milk breastfeeding

INTERVENTIONS:
Other: InFat™ based infant formula — high sn-2 palmitic acid oil based infant formula
  Other Names: high sn-2 palmitic acid; structured triglyceride
  Arms: InFat group
Other: Standard vegetable oil based infant formula — standard vegetable oil based infant formula
  Other Names: standard vegetable oil
  Arms: Control group

SUMMARY:
The purpose of this study is to determine the effect of infant formula with high percentage of palmitic acid at the sn-2 position (InFat™) on improving fat absorption and general gastrointestinal tolerance in Chinese formula-fed term infants.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy of infant formula with high percentage of palmitic acid at the sn-2 position (InFat™) as compared to standard vegetable oil based infant formula on general gastrointestinal tolerance and fat absorption, reducing calcium soaps formation and stool hardness in Chinese formula-fed term infants.

ELIGIBILITY:
Inclusion Criteria:

* Parental/legal guardian written informed consent;
* The mother had unequivocally decided not to breast-feed (for formula fed infants) or to breastfeed (for human milk fed infants).
* Term infant of Chinese origin born at 37-42 gestation weeks
* Birth weight appropriate for gestational age (AGA), 2500-4000grams
* The infant is apparently healthy at birth and entry of study.

Exclusion Criteria:

* Adverse maternal, fetal or infant medical history that can potentially affect efficacy parameters, tolerance, growth and/or development
* The infant is not a singleton newborn

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Soaped and total fatty acids content in infant's stool samples collected at the age of 6 weeks and measured by stool biochemistry analysis | 6 postnatal weeks

SECONDARY OUTCOMES:
Anthropometric parameters: body length, body weight, and head circumferences at each visit | Baseline, 6, 12 and 24 postnatal weeks
Dietary, stool consistency and well being recorded by 3 day questionnaires | 6, 12 and 24 postnatal weeks
Number of participants with adverse events and concomitant medications as a measure of safety and tolerability | Baseline, 6,12 and 24 postnatal weeks
Bone speed of sound measured by ultrasonic device at each visit | Baseline, 6,12 and 24 postnatal weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xu Chundix, Prof., Principal Investigator — Ruijin Hospital
Locations (1):
- Rui Jin Hospital - Shanghai Jiao Tong University School of Medicine, Shanghai, China

REFERENCES:
- [Derived] Bar-Yoseph F, Lifshitz Y, Cohen T, Malard P, Xu C. SN2-Palmitate Reduces Fatty Acid Excretion in Chinese Formula-fed Infants. J Pediatr Gastroenterol Nutr. 2016 Feb;62(2):341-7. doi: 10.1097/MPG.0000000000000971. PMID 26334255